CLINICAL TRIAL: NCT06627023
Title: 3D Analysis of PERI-IMPLANT SOFT TISSUE After Dental Implant Placement with CONICAL and BUTT-JOINT Connection: a 12-Month Randomized Control Trial
Brief Title: 3D Analysis of Peri-implant Soft Tissue with Two Different Connection Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alexey Unkovskiy, MD PhD, Priv.-Doz. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA4_111_24
Record Dates: First submitted 2024-09-28; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Tooth Loss
Keywords: Dental Implants, Implant-Abutment Connection Types, Conical Connection, Butt-Joint Connection, Peri-Implant Soft Tissue, Digital Monitoring
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Intervention Model Description: Example:
  This study uses a parallel-group design, where patients are randomly assigned to either a group with conical connection or a group with butt-joint connection. Soft tissue changes are digitally monitored over a 12-month period.
Who Masked: Investigator
Masking Description: In this study, the primary investigator was informed about the type of implant connection, while the second operator and the patients were not aware of the prosthetic material. No other parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 19 Patients Received Implants with Conical Connections (Active Comparator): Thirty eight patients were enrolled and randomly assigned to receive implants with conical connection. For the first arm 19 patients received implants with conical connections. A standard healing abutment was placed after 6 months for two weeks. The definitive screw-retained crowns were manufactured digitally and delivered afterwards. The soft tissue changes were traced till 12 months post-op
  Interventions: Device: Implant Placement with Conical or Butt-Joint Connection
- 19 Patients Received Implants with Butt-Joint Connections (Active Comparator): Thirty eight patients were enrolled and randomly assigned to receive implants with butt-joint connection. For the first arm 19 patients received implants with conical connections. A standard healing abutment was placed after 6 months for two weeks. The definitive screw-retained crowns were manufactured digitally and delivered afterwards. The soft tissue changes were traced till 12 months post-op
  Interventions: Device: Implant Placement with Conical or Butt-Joint Connection

INTERVENTIONS:
Device: Implant Placement with Conical or Butt-Joint Connection — Thirty eight patients were enrolled in the study and received randomly allocated implants with conical and butt-joint implant-abutment connection type. A standard healing abutment was placed after 6 months for two weeks. The definitive screw retained crowns were manufactured in a digital workflow. The soft tissue profile was digitized using IOS on following stages: pre-op, post-op: immediately, two, 7 and 14 days, pre-exposure, immediately after exposure, two weeks after exposure (pre-delivery), immediately after crown delivery, 6 and 12 months post-op.

SUMMARY:
Objectives: assessment of dimensional soft tissues change after single tooth gap implantation with a closed healing approach and using conical and butt-joint implant-abutment connection type.

Material and Methods: forty patients were enrolled in the study and received randomly allocated implants with conical and butt-joint implant-abutment connection type. A standard healing abutment was placed after 6 months for two weeks. The definitive screw retained crowns were manufactured in a digital workflow. The soft tissue profile was digitized using IOS on following stages: pre-op, immediately, two, 7 and 14 days post-op, pre-exposure, immediately after exposure, two weeks after exposure (pre-delivery), immediately after crown delivery, 6 and 12 months after delivery. The intraoral scans were matched in the metrology software (Geomagic Control X). The mean maximum and mean average differences in mm were gathered to assess the soft tissues change. Various anamnesis parameters have been taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a single tooth gap, completion of conservative and periodontal treatments, diagnostic preoperative models, and a recent panoramic radiograph not older than 6 months.

Exclusion Criteria:

* Abnormal jaw anatomy, insufficient bone volume, bone conditions (e.g., cysts, tumors), oral mucosa abnormalities (e.g., lesions, diseases), untreated periodontal disease, acute inflammation, pregnancy, temporary medication contraindications, psychological issues (e.g., substance abuse), poor compliance, and general medical contraindications.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Linear changes of soft tissue in mm | Assessment at pre-op, immediately post-op, 2 days, 7 days, 14 days, pre-exposure, post-exposure, pre-delivery, immediately after crown delivery, 6 months, and 12 months.
  The primary outcome measure is the change in peri-implant soft tissue profile, quantified in millimeters, assessed at various stages post-op. This includes measurements taken at pre-operative, immediately post-operative, 2 days, 7 days, 14 days, pre-exposure, post-exposure, pre-delivery, immediately after crown delivery, and at 6 and 12 months after delivery.

SECONDARY OUTCOMES:
Influence of anamnestic parameters | 12 months
  For all enrolled patients a detailed medical history was collected, including following parameters: sex, region, brushing, mouth rinsing, flossing, alcohol consumption, stress, periodontitis therapy, gingival biotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to confidentiality concerns and the need to protect patient privacy.

REFERENCES:
- [Background] 1. Warreth, A., et al., Dental implants and single implant-supported restorations. J Ir Dent Assoc, 2013. 59(1): p. 32-43. 2. Wang, Y., et al., Patient satisfaction and oral health-related quality of life 10 years after implant placement. BMC Oral Health, 2021. 21(1). 3. Hebel, K., R. Gajjar, and T. Hofstede, Single-tooth replacement: bridge vs. implant-supported restoration. J Can Dent Assoc, 2000. 66(8): p. 435-8. 4. Gomez-Meda, R., J. Esquivel, and M.B. Blatz, The esthetic biological contour concept for implant restoration emergence profile design. Journal of Esthetic and Restorative Dentistry, 2021. 33(1): p. 173-184. 5. Kadkhodazadeh, M., et al., Timing of soft tissue management around dental implants: a suggested protocol. Gen Dent, 2017. 65(3): p. 50-56. 6. Siegenthaler, M., et al., Anterior implant restorations with a convex emergence profile increase the frequency of recession: 12-month results of a randomized controlled clinical trial. Journal of Clinical Periodontology, 2022. 49(11): p. 1145-1157. 7. Tavelli, L., et al., Peri-implant soft tissue phenotype modification and its impact on peri-implant health: A systematic review and network meta-analysis. Journal of Periodontology, 2021. 92(1): p. 21-44. 8. Gomez-Meda, R., J. Esquivel, and M.B. Blatz, The esthetic biological contour concept for implant restoration emergence profile design. J Esthet Restor Dent, 2021. 33(1): p. 173-184. 9. Luo, R.M., et al., Soft-Tissue Grafting Solutions. Dent Clin North Am, 2020. 64(2): p. 435-451. 10. Deeb, G.R. and J.G. Deeb, Soft Tissue Grafting Around Teeth and Implants. Oral Maxillofac Surg Clin North Am, 2015. 27(3): p. 425-48. 11. Jepsen, S., et al., Primary prevention of peri-implantitis: Managing peri-implant mucositis. Journal of Clinical Periodontology, 2015. 42: p. S152-S157. 12. Laleman, I. and F. Lambert, Implant connection and abutment selection as a predisposing and/or precipitating factor for peri-implant diseases: A review. Clin Implant Dent Relat Res, 202
- [Background] 15. Ruales-Carrera, E., et al., Peri-implant tissue management after immediate implant placement using a customized healing abutment. J Esthet Restor Dent, 2019. 31(6): p. 533-541. 16. Thoma, D.S., et al., Effects of soft tissue augmentation procedures on peri-implant health or disease: A systematic review and meta-analysis. Clin Oral Implants Res, 2018. 29 Suppl 15: p. 32-49. 17. Thoma, D.S., et al., Efficacy of soft tissue augmentation around dental implants and in partially edentulous areas: a systematic review. J Clin Periodontol, 2014. 41 Suppl 15: p. S77-91. 18. Ramanauskaite, A., et al., Three-dimensional changes of a porcine collagen matrix and free gingival grafts for soft tissue augmentation to increase the width of keratinized tissue around dental implants: a randomized controlled clinical study. Int J Implant Dent, 2023. 9(1): p. 13. 19. Mancini, L., et al., 3D surface defect map for characterising the buccolingual profile of peri-implant tissues. Int J Oral Implantol (Berl), 2023. 16(2): p. 105-113. 20. Buda, M., M. Bratos, and J.A. Sorensen, Accuracy of 3-dimensional computer-aided manufactured single-tooth implant definitive casts. J Prosthet Dent, 2018. 120(6): p. 913-918. 21. Kernen, F., et al., A review of virtual planning software for guided implant surgery - data import and visualization, drill guide design and manufacturing. BMC Oral Health, 2020. 20(1): p. 251. 22. Poppolo Deus, F. and A. Ouanounou, Chlorhexidine in Dentistry: Pharmacology, Uses, and Adverse Effects. Int Dent J, 2022. 72(3): p. 269-277. 23. Pesce, P., et al., Systematic review of some prosthetic risk factors for periimplantitis. J Prosthet Dent, 2015. 114(3): p. 346-50. 24. AlQarawi, F.K., et al., Microleakage and Bacterial Adhesion with Three Restorative Materials Used to Seal Screw-access Channels of Implant Abutments: An In vitro Study. Saudi J Med Med Sci, 2021. 9(3): p. 241-247. 25. Amornvit, P., D. Rokaya, and S. Sanohkan, Comparison of Accuracy of Current Ten Intraoral S
- [Background] Farronato, D., et al., Behavior of Soft Tissue around Platform-Switched Implants and Non-Platform-Switched Implants: A Comparative Three-Year Clinical Study. J Clin Med, 2021. 10(13). 31. Rodrigues, V.V.M., et al., Is the clinical performance of internal conical connection better than internal non-conical connection for implant-supported restorations? A systematic review with meta-analysis of randomized controlled trials. J Prosthodont, 2023. 32(5): p. 382-391. 32. López-Marí, L., et al., Implant platform switching concept: an updated review. Med Oral Patol Oral Cir Bucal, 2009. 14(9): p. e450-4. 33. Schmitt, C.M., et al., Performance of conical abutment (Morse Taper) connection implants: a systematic review. J Biomed Mater Res A, 2014. 102(2): p. 552-74. 34. Gupta, S., et al., Platform switching technique and crestal bone loss around the dental implants: A systematic review. Ann Afr Med, 2019. 18(1): p. 1-6. 35. Ackermann, K.L., et al., Clinical and patient-reported outcome of implant restorations with internal conical connection in daily dental practices: prospective observational multicenter trial with up to 7-year follow-up. Int J Implant Dent, 2020. 6(1): p. 14. 36. Ramanauskaite, A. and R. Sader, Esthetic complications in implant dentistry. Periodontol 2000, 2022. 88(1): p. 73-85. 37. Chow, Y.C. and H.L. Wang, Factors and techniques influencing peri-implant papillae. Implant Dent, 2010. 19(3): p. 208-19. 38. Stefanini, M., et al., Peri-implant Papillae Reconstruction at an Esthetically Failing Implant. Int J Periodontics Restorative Dent, 2020. 40(2): p. 213-222. 39. Smukler, H., F. Castellucci, and D. Capri, The role of the implant housing in obtaining aesthetics: generation of peri-implant gingivae and papillae--Part 1. Pract Proced Aesthet Dent, 2003. 15(2): p. 141-9; quiz 150.